CLINICAL TRIAL: NCT00467376
Title: 12-week, Multicenter, Controlled, Open, 3:1 Randomized, Parallel Clinical Trial Comparing Insulin Glulisine With Regular Human Insulin (Insulin Lispro) Injected Subcutaneously in Subjects With Type 1 or 2 Diabetes Mellitus Also Using Lantus (Insulin Glargine)
Brief Title: Insulin Glulisine, Insulin Lispro and Insulin Glargine in Type 1 or 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_00348
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin glulisine; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Administration of Insulin Glulisine
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Glargine
- 2 (Active Comparator): Administration of Lispro
  Interventions: Drug: Lispro; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glulisine — 3 times a day before each meal
  Arms: 1
Drug: Lispro — 3 times a day before each meal
  Arms: 2
Drug: Insulin Glargine — once daily

SUMMARY:
Primary:

* To compare the efficacy and safety of Insulin Glulisine to Insulin Lispro in subjects with type 1 or type 2 diabetes mellitus.
* To compare the frequency of hypoglycemia of Insulin Glulisine to Insulin Lispro.

Secondary:

* To compare Insulin Glulisine to Insulin Lispro in terms of the change in HbA1c at weeks 12, blood glucose parameters, insulin doses and treatment satisfaction in subjects with type 1 or type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetic patients
* Measure HbA1c 6.5% to 11.0% at visit 1
* More than 3 months of continuous insulin treatment immediately prior to study entry

Exclusion Criteria:

* Pregnant women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Hypoglycemic episodes | From the beginning to end of the study
Change in HbA1c | From baseline to endpoint
Adverse events | From the beginning to the end of study

SECONDARY OUTCOMES:
Change in HbA1c | From baseline to weeks 12
blood glucose parameters, hypoglycemic episodes and dosage of the mealtime and Lantus. | from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jing Fu, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Beijing, China